CLINICAL TRIAL: NCT00532285
Title: Phase II Study of Primary Paclitaxel Plus Gemcitabine in Patients With Stage II and III Breast Cancer
Brief Title: Primary Paclitaxel Plus Gemcitabine in Patients With Stage II and III Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: CENTER FOR BREAST CANCER, NATIONAL CANCER CENTER
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-05-150
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel/Gemcitabine (Experimental): paclitaxel 80 mg/m2 (day 1, 8) and gemcitabine 1200 mg/m2 (day1, 8) every 3 weeks, 4 cycles
  Interventions: Drug: Paclitaxel/Gemcitabine

INTERVENTIONS:
Drug: Paclitaxel/Gemcitabine — Treatment will be delivered in the outpatient setting. Each three-week cycle consists of paclitaxel 80 mg/m2 (day 1, 8) and gemcitabine 1200 mg/m2 (day1, 8).Patients will receive four cycles of therapy unless there is any evidence of no response (SD or PD) or unacceptable toxicity defined as unpredictable, irreversible, or Grade 4, or noncompliance by patient with protocol requirements.
  Other Names: Paclitaxel; Gemzar

SUMMARY:
This is an open labeled phase II single arm trial. The patients with clinical stage II and III will undergo core-needle biopsy of breast tumor for histologic diagnosis, immunohistochemical studies for estrogen receptor (ER), progesterone receptor(PR), HER-2/neu and others. PET or ultrasound results will determine the positivity of lymph node metastasis.

DETAILED DESCRIPTION:
Patients will be treated as follows:

PG x 4®operation®AC x 4®radiation ± tamoxifen/AI(postmenopausal)

Intravenous infusion of Paclitaxel 80 mg/m2, over 60 min, on D1 and D8 Followed by intravenous infusion of Gemcitabine 1200 mg/m2, over 30 min, on D1 and D8

The cycle repeats every 3 weeks for 4 times. Premedication includes antiemetics, dexamethasone, famotidine, pheniramine as routinely given.

After the operation, standard adjuvant chemotherapy (doxorubicin 60 mg/m2, cyclophosphamide 600 mg/m2, every 3 weeks x 4 cycles) will be given.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically confirmed and newly diagnosed breast cancer: node-positive stage IIA and any stage IIB, III. PET results will determine node positivity. If PET was not utilized, sonographically positive node should be confirmed cytologically by fine needle aspiration.
* No prior hormonal, chemotherapy or radiotherapy is allowed.
* No breast operation other than biopsy to make diagnosis is allowed.
* Age: 18-years and older, not pregnant pre-, and postmenopausal women with good performance status (ECOG 0-1)
* Adequate hematopoietic function: Absolute granulocyte count ³1500/mm3, platelet ³100,000/mm3, Hemoglobin ³ 10 g/mm3
* Adequate renal function: Serum creatinine £ 1.5 mg/dl
* Adequate hepatic function: total bilirubin: £ 1.5 mg/dl, AST/ALT: £ two times normal, Alkaline phosphatase: £ two times normal
* Adequate cardiac function: normal or nonspecific EKG taken within 1 mo of enrollment
* Adequate mental function to understand and sign the consent

Exclusion Criteria:

* Patients who received hormonal, chemotherapy or radiotherapy for breast cancer
* Patients who underwent surgery for breast cancer
* Patients with node-negative stage IIA breast cancer
* Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-09; Primary Completion 2006-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical and pathologic responses to preoperative administration of Paclitaxel/Gemcitabine (PG) | two years

SECONDARY OUTCOMES:
To assess breast conserving rate To evaluate the disease free survival (DFS) and overall survival (OS) of patients who received preoperatively PG To investigate the toxicity profiles of PG | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, MD, PhD, Principal Investigator — National Cancer Center